Exploring the Effect of Rumination-Focused Cognitive Behavior Therapy on Depressive Symptoms in Patients with Schizophrenia: A Randomized Controlled Trial

NCT04442893 31 MAY 2019 (IRB1080909-01)

## **Background**

Depression is one of the core symptoms in schizophrenic patients. Studies have shown that schizophrenic patients have a higher suicidal thought than the general population was due to depressive symptoms. Thus, the impact of depressive symptoms in schizophrenic patients demands significant attention.

### Aim

The aim of this study was to examine the impact of rumination-focused cognitive behaviour therapy (RFCBT) on depressive symptoms, responses to rumination, personal stigma and hope in patients with Schizophrenia.

# Design

The study was a randomized, controlled, single-blind study; non-probability sampling was used to recruit participants. The recovery ward of a specialized psychiatric hospital in northern Taiwan was used for field study. The second author, who did not contact the study subjects, used Random Allocation Software Vision 2.0 (Saghaei, 2004) to perform 4-block randomization of the participants [20]. In the experimental group (EG), RFCBT was conducted in groups, and routine nursing care was maintained. The control group (CG) received health education in groups. A structured questionnaire, administered by 3 nursing staff members who were not researchers, was used for data collection; the questionnaire was administered 3 times: before the intervention (T0), after the intervention (T1), and 3 months after the intervention (T2).

#### Methods

The study was conducted in seven wards of a psychiatric center in northern Taiwan. Eighty-five participants with schizophrenia were enrolled. The group allocation was conducted using a block randomization software program. The experimental group (n = 44) was provided with a 6-session RFCBT program in 12 weeks (at least 90 minutes a session biweekly), while the Control group (n = 41) received a 6-session psychosocial education program in 12 weeks (at least 60 minutes biweekly). All

data collection took place between July 2019 and March 2020. A structured questionnaire were used to collect data on demographic data, Beck Depression Inventory II(BDI-II), Chinese Response Style Questionnaire-short form revised(CRSQ-10), the Internalized Stigma of Mental Illness Scale(ISMIS) and Herth Hope Index Chinese Version(HHI) at baseline, post-intervention and 3-month follow-up.

## **Statistical Analysis Plan**

This study employed IBM SPSS Statistics 24.0 to analyze the collected data for a two-tailed test with a 0.05 significance level. The descriptive statistics included mean, standard deviation, frequency, and percentages; the inferential statistics included  $\chi 2$  test, independent t-test and the generalized estimating equation (GEE) were employed to explore the effect of RFCBT on improving depression-related symptoms, rumination response, self-stigma and hope after controlling demographic data.